CLINICAL TRIAL: NCT05101161
Title: Neurofeedback Using Implanted Deep Brain Stimulation Electrodes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Responsible Party: Principal Investigator, Oliver Bichsel, Principal Investigator, ETH Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NF-DBS
Record Dates: First submitted 2021-09-23; First posted 2021-11-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Epilepsy; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Epilepsy; Essential Tremor | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bidirectional Neurofeedback (Experimental)
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback — Modulating brain oscillations based on visual neurofeedback

SUMMARY:
Deep brain stimulation (DBS) has become a gold-standard symptomatic treatment option for Parkinson's disease (PD) and is also explored for a variety of other neurological disorders. The implantation of electrodes into deep brain areas has not only enabled the application of electrical stimuli, but has also provided researchers and clinicians with an unprecedented window to investigate aberrant neuronal activity right at the core of pathological brain circuits. Local field potentials (LFP) have already been readily investigated through externalised DBS electrode wires prior to internalisation and connection to an implantable neurostimulator. In the case of PD, motor symptoms have been evidenced to correlate with exaggerated beta oscillatory activity (13-35 Hz) in the LFP recorded from the subthalamic nucleus (STN). Firstly, beta activity recorded in the STN at rest in patients withdrawn from their medication has been correlated with the Unified Parkinson's Disease Rating Scale (UPDRS) across patients. Secondly, a reduction of signal power in the beta-band was correlated with clinical improvements of motor symptoms. Thirdly, the two main therapeutic strategies, the administration of L-Dopa, and high-frequency DBS both lead to a suppression of beta-synchronicity in the STN. Furthermore, beta-oscillations show fast and movement-dependent modulation over time and can serve as a biomarker and feedback signal to control the delivery of DBS. The investigators recently implemented deep brain electrical neurofeedback to provide real-time visual neurofeedback of pathological STN oscillations through externalised DBS electrodes and showed that PD patients were able to volitionally control and reduce subthalamic activity within a single 1 hour session. Moreover, neurofeedback-learnt strategies accelerated movements and could be retained in the short- and mid-term. Only recently, a newly developed neurostimulator, the Percept™ PC (Medtronic Neurological Division, Minneapolis, MN, USA), has been clinically approved, which can not only apply electrical impulses, but also enable the measurement and transmission of brain activity. This neurostimulator is now the first choice for implantations at the University Hospital Zurich and is used for a variety of neurological disorders. The investigators' goal is to investigate whether neurofeedback through a fully implanted deep brain stimulation device is possible and can lead to a better control of pathological oscillations as well as symptom mitigation. Having shown that endogenous control over deep brain oscillations is possible, the investigators will also test this novel therapeutic approach for pathologies other than PD that are also treated with DBS. Neurofeedback using implanted DBS electrodes will have the advantage of enabling longer and multiple-day training sessions, which the investigators hypothesise to have a larger impact on control over pathological deep brain oscillations and neurological symptoms, as such a fully implanted neurofeedback system no longer requires the externalisation of DBS wires and is as such no longer limited to the first two days after electrode implantation. All in all, the investigators will not exceed a total streaming time of 7 hours per patients (7 d of battery time), which the investigators deem justifiable with respect to a battery life of > 5 years. This proposed research is highly significant as it will help our understanding of various neurological diseases that are highly prevalent in society (PD being, for instance, the second most common neurodegenerative disorder after Alzheimer's disease) and might culminate in novel, endogenous treatment strategies. The overall risk for patients is minimal to non-existent, as stimulation parameters are unaffected and the intended changes in brain activity are self-induced while DBS stimulation is off.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing clinically indicated implantation of a Percept™ PC neurostimulator, age ≥ 18 years as well as planned hospitalisation of ≥ 3 days after operation

Exclusion Criteria:

minimal prognosticated survival of less than 1 year, reduced state of consciousness (i. e. Glasgow Coma Scale < 15), inability to communicate (in terms of hearing, seeing, speaking and understanding), other significant concomitant diseases (e. g. cardiovascular disease, infectious disease, isolation), inability to follow procedures, insufficient knowledge of project language, inability to give consent and unlikeliness to follow protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Amount of endogenous neuromodulation (difference in oscillatory power) | 60 Minutes
  The investigators will assess the amount of endogenous modulation of the neurofeedback parameter as compared to a baseline state ('rest') as well as in a bidirectional neurofeedback design (upregulation vs. downregulation). Local field potentials are measured (LFP-recording; physiological parameter; for Parkinson patients the beta-frequencies will be assessed during the study period) using already implanted deep brain stimulation electrodes (Medtronic DBS electrodes) and used to compute the neurofeedback parameter. The amount of endogenous neuromodulation is determined as the difference of power of neuronal oscillations between two conditions [unit of measure: %-difference in power of deep brain neuronal oscillations].

SECONDARY OUTCOMES:
performance in motor activity tasks | 60 min
  The investigators will assess the 'performance in motor activity tasks' (= name of the measurement) using the measurement tools of wearable inertial measurement units (IMUs) and motion detectors. The following units of measure (physiological parameters) could be extracted from the recorded data: speed of movement, smoothness of movement, extent of movement.
transfer of neurofeedback-learnt strategies | 60 min
  The investigators will assess the amount of endogenous modulation of the neurofeedback parameter as compared to a baseline state ('rest') as well as in a bidirectional neurofeedback design (upregulation vs. downregulation) in the ABSENCE of active neurofeedback. Local field potentials are measured (LFP-recording; physiological parameter; for Parkinson patients the beta-frequencies will be assessed during the study period) using already implanted deep brain stimulation electrodes (Medtronic DBS electrodes) and used to compute the neurofeedback parameter. The amount of endogenous neuromodulation is determined as the difference of power of neuronal oscillations between two conditions [unit of measure: %-difference in power of deep brain neuronal oscillations].
agency as measured on a visual scale (1-10) | 60 min
  the subjectively perceived ability to control deep brain oscillatory activity. Patients will be asked to indicate the perceived ability (agency) to control the neurofeedback parameter on a visual scale from 0 (no control) to 10 (perfect control).

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Bichsel, MD, MSc ETH, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided